CLINICAL TRIAL: NCT04530279
Title: Accordance of Clinical Assessment of Burn Depth and %TBSA Between Referring Hospitals and the National Norwegian Burn Centre
Brief Title: Clinical Assessment of Burns in Norway
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/1627, Rek-Vest
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Burns
Keywords: clinical assessment; TBSA; national burn centre
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Referring hospital: Burn assessments performed in referring hospitals
  Interventions: Procedure: Clinical assessment
- Burn centre: Burn assessments performed in the national burn centre
  Interventions: Procedure: Clinical assessment

INTERVENTIONS:
Procedure: Clinical assessment — Clinical assessment of burn depth and the percentage of total body surface area (TBSA) burnt with any method

SUMMARY:
Clinical assessment of burn depth and area can be challenging even for experienced surgeons. Still, the assessment is fundamental for the treatment, as it determines the fluid treatment and indication for escharotomy and need for referral to a burn centre.There are few studies comparing the initial evaluation of burn depth and surface with that of a specialist burn centre. The aim of this study was to make such a comparison for a cohort of patients admitted to a specialist burn centre during one year.The cohort was defined as patients transferred to the burn unit at Haukeland university hospital during 2014.

ELIGIBILITY:
Inclusion Criteria:

* Patients transferred to the burn unit at Haukeland university hospital during 2014

Exclusion Criteria:

* Readmissions
* Patients transported to Haukeland directly from the site of the accident

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The cohort was defined as patients transferred to the burn unit at Haukeland university hospital during 2014.The incidence of burns in Norway is 15.5 /100 000/ year (pop.
  5.2 mill), and 70-100 patients a year is treated at the national burn centre. The
  Australian and New Zealand Burn Association (ANZBA) referral criteria are used:
  * Burns > 10% Total Body Surface Area (TBSA)
  * Burns > 5% TBSA in children
  * Full Thickness burns > 5% TBSA
  * Burns of Special Areas - Face, Hands, Feet, Genitalia, Perineum, Major Joints and circumferential limb or chest burns
  * Burns with inhalation injury
  * Electrical burns
  * Chemical burns
  * Burns with pre-existing illness
  * Burns associated with major trauma
  * Burns at the extremes of age - young children and the elderly
  * Burn injury in pregnant women
  * Non-accidental burns
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Burn depth | 1 year
  Burn depth measured with any described clinical method.Clinical assessment of depth is a subjective evaluation based on visual and tactile characteristics, that is, wound appearance, capillary refill and wound sensibility to touch and pin prick.
The percentage of total body surface area (TBSA) burnt | 1 year
  TBSA measured with any described clinical method, for example, Wallace's Rule of Nines, Lund and Browder charts, and Palmar Surface Measurement ('rule of palm')

CONTACTS AND LOCATIONS:
Overall Officials: Ragnvald L Brekke, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No